CLINICAL TRIAL: NCT01798082
Title: Effect of a Decision Aid on Decision Making for the Treatment of Pelvic Organ Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Hema Brazell, Principal Investigator, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: BRAZ003846HU; 333590
Record Dates: First submitted 2013-02-20; First posted 2013-02-25 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Decisional Conflict

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard counseling (No Intervention)
- Standard counseling, pelvic organ prolapse decision aid (Experimental): In addition to standard counseling at the time of the initial new patient visit, the patients randomized to the experimental arm will recieve a pelvic organ prolapse decision aid prior to their initial visit.
  Interventions: Other: Pelvic organ prolapse decision aid

INTERVENTIONS:
Other: Pelvic organ prolapse decision aid
  Arms: Standard counseling, pelvic organ prolapse decision aid

SUMMARY:
Pelvic organ prolapse is a common condition that affects millions of women every year. There are many options for treatment and it can be difficult to make a decision as how best to proceed. Previous studies have shown that decisional aids (DAs) may improve knowledge, physician-patient communication, decisional conflict, and patient satisfaction. However, no study has evaluated the role of a decisional aid among women presenting for evaluation and management of prolapse. We would like to determine if a decision aid for prolapse decreases the amount of decisional conflict women face when choosing a plan of care.

We hypothesize that there will be a difference in the level/amount of decisional conflict between women who receive a DA and those who do not. Specifically, we anticipate that women randomized to receiving standard counseling and a DA with have less decisional conflict than the cohort receiving standard counseling alone.

DETAILED DESCRIPTION:
Women scheduled for the evaluation and management of pelvic organ prolapse at Hartford Hospital will be contacted via telephone prior to the initial consultation visit to ascertain interest for this study. If they are interested, they will be randomized to one of two groups: those that receive a DA and those that do not.

This study requires you to answer some questions about the information packet you received in the mail. We routinely send a packet to all of our new patients. Half of the participants received a decision aid to supplement their information packet and the other half received our routine informational packet. You will be asked to complete a set of 2 questionnaires. It will take less than 10 minutes to complete these questions.

All data will be extracted and used by only the investigators on this study. The data will be stored on a restricted-access network drive and results will be reported in aggregate and no personal health history will be disclosed. Our primary outcome for this analysis is decisional conflict differences in those who receive a DA and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Female
* ≥18 years old
* Scheduled for consultation visit for pelvic organ prolapse of any type (cystocele, rectocele, enterocele, uterine prolapse, and/or uterovaginal prolapse)

Exclusion Criteria:

* <18 years old
* Non-English speaking
* Any patient who declines, or expresses unwillingness to being contacted for participation in the study
* Planned concomitant non-gynecologic procedure
* Established patient in the practice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Difference in decisional conflict | 1 year
  The primary outcome for this analysis is decisional conflict differences in those who receive a DA and those who do not. The investigators will administer the 16-item traditional Decisional Conflict Scale (DCS). The DCS comprises 3 subscales: decision uncertainty, factors contributing to uncertainty, and perceived effective decision making. The investigators will use the statement format of this scale in which patients respond to a series of Likert-scale statements using response categories of strongly agree, agree, neither agree nor disagree, disagree, or strongly disagree, which are scored as 0-4, respectively, and added. Based on previous research, scores will be tabulated and patients will be grouped as either having "high level of decisional conflict" versus "low level of decisional conflict."
  Values will be assessed for normality and compared between groups (i.e. those receiving the DA versus those who did not).

SECONDARY OUTCOMES:
Number of patients who choose surgery over conservative management | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hema Brazell, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States